CLINICAL TRIAL: NCT00561106
Title: Treatment Bell´s Palsy: Prednisone vs Prednisone Valacyclovir
Brief Title: Prednisone-Placebo vs Prednisone-Valacyclovir in Bell´s Palsy
Acronym: PVBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de la Republica (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HC 6-8-02
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Bell´s Palsy
Keywords: Bell´s palsy; prednisone; valacyclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: prednisone- valacyclovir
- 2 (Placebo Comparator)
  Interventions: Drug: prednisone-placebo

INTERVENTIONS:
Drug: prednisone- valacyclovir — prednisone, a dose of 1 mg/kg body weight was given daily for 7 days. The treatment was tapered over the next 14 days. Those taking valacyclovir received 1000 mg in two daily doses for 7 days.
  Arms: 1
Drug: prednisone-placebo — prednisone, a dose of 1 mg/kg body weight was given daily for 7 days
  Arms: 2

SUMMARY:
Since steroids carry a moderate beneficial effect in Bell's palsy, and to address this question, valacyclovir was added to prednisone for the treatment of this condition.

DETAILED DESCRIPTION:
Between December 2002 and December 2003, a total of 52 subjects with BP were evaluated, 42 fulfilled the inclusion criteria and entered the study, 1 patient was lost to follow-up after the first visit, leaving a total of 41 patients with complete clinical follow-up.

To be included in the study, patients had to be evaluated within the first 72 hours and could have no contraindications to steroid or valacyclovir therapy.

Patients were randomly assigned to either the prednisone-valacyclovir (group 1) or the prednisone-placebo group (group 2) Among the 41 patients completing the study, 19 pertenecian al group 1 and 21 group 2 Both groups received prednisone, a dose of 1 mg/kg body weight was given daily for 7 days (one single dose after breakfast). The treatment was tapered over the next 14 days. Those taking valacyclovir received 1000 mg in two daily doses for 7 days. All subjects were instructed about eye protection and lubrication were followed at regular intervals until recovery or for a minimum period of 3 months. Follow-up included examination at 1, 2, 4, 8 and 12 weeks after the first visit. Patients with incomplete recovery at 3 months were controlled until complete recovery or stabilization of the paralysis. All subjects were evaluated for laboratories parameters. Routine blood count, blood sugar, and liver function tests were performed at first visit.

There were no severe side effects attributable to the valacyclovir-prednisone treatment in this study.

Informed consent was obtained from all patients. Facial nerve function was assessed using the facial grading system (FGS) The scale used provides a quantitative score with three components; resting symmetry, symmetry of voluntary movement and synkinesis and a composite score was obtained.

Student's t-test was employed for quantitative….variables. Comparison of treatment results between both groups was performed by….means of an analysis of variance (ANOVA) test of two ways (therapy and time).

All statistical tests were considered received the same level of significance (P = 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Patients with Bell´s palsy evaluated within the first 72 hours.

Exclusion Criteria:

* Peptic ulcer
* Tuberculosis
* Moderate or severe diabetes
* Moderate or severe hypertension
* Glaucoma
* Manifest cardiac disease
* Psychosis
* Renal or hepatic dysfunction, and
* Pregnancy.

Ages: 14 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2002-12; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
The following parameters were used to evaluate the final result: grade of recovery, and sequelae.Facial nerve function was assessed using the facial grading system (FGS) Normal recovery was defined as the return of facial function to FGS 90 or more. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Vazquez, Dr., Principal Investigator — Hospital de Clinicas Facultad de Medicina Universidad de la Republica
Locations (1):
- Hospital de clinicas, Montevideo, Montevideo Department, Uruguay